CLINICAL TRIAL: NCT04433975
Title: Psychosocial Pain Management to Improve Opioid Use Disorder Treatment Outcomes: A Randomized Controlled Trial
Brief Title: Psychosocial Pain Management to Improve Opioid Use Disorder Treatment Outcomes
Acronym: Persist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark A. Ilgen, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HUM00166747; R33AT010106 (NIH); R01AT010797 (NIH)
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Results first posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder; Medication Assisted Treatment; Chronic Pain
Keywords: Psychosocial Pain Management; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial Pain Management (PPMI) (Experimental): Eight Cognitive Behavioral Therapy-based individual telephone or video therapy sessions with research study therapist.
  Interventions: Behavioral: Psychosocial Pain Management (PPMI)
- Enhanced Usual Care (EUC) (Active Comparator): Two individual telephone educational sessions with research study therapist.
  Interventions: Behavioral: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: Psychosocial Pain Management (PPMI) — The main theme of the treatment is to provide participants with new ways of thinking and coping skills related to managing pain and opioid use in order to increase the likelihood the participant may remain in buprenorphine treatment.
  Arms: Psychosocial Pain Management (PPMI)
Behavioral: Enhanced Usual Care (EUC) — The EUC condition is designed to match the PPMI condition in terms of the non-specific aspects of receiving support for pain, substance use, and receiving monitoring of buprenorphine adherence.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The purpose of this research study is to look at the effect of programs aimed at helping people manage chronic pain and medication treatment. The program sessions focus on educational information and strategies for pain and medication management. The researchers enroll people who have chronic pain and have recently begun buprenorphine treatment to see if participants could benefit from these programs. This research study will help the researchers learn how to improve current therapies for pain and medication management.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of an opioid use disorders (OUD) within the past 12 months;
* started buprenorphine (the term we use to refer to all buprenorphine products including buprenorphine/naloxone) treatment within the past 6 months
* at least moderate or greater self-reported pain on average over the past 3 months;
* regular and consistent access to a telephone and willingness to use the phone for study sessions.

Exclusion Criteria:

* buprenorphine medication prescribed in the form of a monthly injection and/or a transdermal patch
* self-reported pregnancy at the time of study enrollment
* currently living outside of the United States

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2025-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lin, M.D., M.S., Principal Investigator — University of Michigan; Mark Ilgen, Ph.D., Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Veterans Affair Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Michigan Medicine, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ilgen M, Blow F, Piette JD, Goldstick J, Lewis M, Priest W, Matharu H, Bourgoise M, Young C, Ashe D, Price A, Lin LA. The psychosocial pain management to improve opioid use disorder treatment outcomes study: Protocol for a randomized controlled trial. Contemp Clin Trials. 2025 Nov;158:108081. doi: 10.1016/j.cct.2025.108081. Epub 2025 Sep 17. PMID 40972890

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IRB approval from the University of Michigan (UM) was obtained in February 2020 with remote recruitment changes approved in June 2020. Several of the recruitment strategies used were in person recruitment at local buprenorphine clinics; posted flyers at community locations; targeted advertising on Facebook, Instagram, and Craigslist; posts on the UMHealthResearch.org page; advertising on websites that target patients in recovery; review of health records at UM and Ann Arbor VA Healthcare System
Period: Completed Baseline and Randomized
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Started | 98 | 102
Completed | 98 | 102
Not Completed | 0 | 0
Period: 1-month Follow Up
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Started | 98 | 102
Completed Interview | 81 | 82
Completed (Completed = number of participants that completed the timepoint survey.) | 76 | 76
Not Completed | 22 | 26
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 21 | 25
Period: 3-month Follow Up
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Started | 97 | 101
Completed Interview | 78 | 84
Completed (Completed = number of participants that completed the timepoint survey.) | 74 | 77
Not Completed | 23 | 24
Not completed — Lost to Follow-up | 20 | 24
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: 6-month Follow Up
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Started | 94 | 101
Completed Interview | 72 | 74
Completed (Completed = number of participants that completed the timepoint survey.) | 70 | 72
Not Completed | 24 | 29
Not completed — Lost to Follow-up | 23 | 28
Not completed — Withdrawal by Subject | 1 | 1
Period: 9-month Follow Up
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Started | 93 | 100
Completed Interview | 69 | 70
Completed (Completed = number of participants that completed the timepoint survey.) | 66 | 63
Not Completed | 27 | 37
Not completed — Lost to Follow-up | 27 | 36
Not completed — Death | 0 | 1
Period: 12-month Follow Up
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Started | 93 | 99
Completed Interview | 68 | 73
Completed (Completed = number of participants that completed the timepoint survey.) | 66 | 68
Not Completed | 27 | 31
Not completed — Lost to Follow-up | 27 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 98 | 102 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.37 (10.79) | 44.68 (10.78) | 43.55 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 41 | 44 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 4 | 12
  Not Hispanic or Latino | 88 | 97 | 185
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 8 | 20
  White | 75 | 90 | 165
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 98 | 102 | 200
Military Status [Count of Participants; unit: Participants] — Self-identified yes/no to "Have you ever been in the United States Armed Forces?"
  Participants | 2 | 5 | 7
Brief Pain Inventory (BPI) Score [Mean (Standard Deviation); unit: units on a scale] — Pain-related functioning will be measured using the pain interference subscale of the Brief Pain Inventory - Short Form (BPI), an 11-point numeric rating scale (0 = no pain/does not interfere, 10 = worst pain imaginable/completely interferes).
  units on a scale | 4.7 (2.2) | 4.8 (2.4) | 4.8 (2.3)
Percent days abstinent [Mean (Standard Deviation); unit: percent] — During the TimeLine Follow Back assessment at baseline, participants reported their daily substance use for the past 6 months. The team calculated the average percentage of days that participants did not use substances within the 6-month period prior to their baseline assessment ((# of days abstinent )/(# of baseline days assessed)*100).
  percent | 51.3 (33.2) | 50.9 (34.0) | 51.1 (33.6)
Numeric Rating Scale (NRS-I) Score [Mean (Standard Deviation); unit: units on a scale] — Pain level will be measured using the Numerical Rating Scale for Pain Intensity (NRS-I), an 11-point numeric rating scale (0 = no pain, 10 = worst pain imaginable).
  units on a scale | 7.43 (1.28) | 7.55 (1.26) | 7.49 (1.28)
Rapid Opioid Dependence Screen (RODS) [Mean (Standard Deviation); unit: units on a scale] — RODS is an 8-item measure based on the DSM criteria that is used to quickly assess opioid dependence among adults. RODS assesses lifetime use of opioids such as heroin, methadone, buprenorphine, oxycontin, and other opioid analgesics, and asks questions measuring physiological, behavioral, and cognitive factors associated with opioid use. RODS uses binary (yes/no) responses that are summed to create the summary measure. Summary scores range from 0 - 8, with "Yes" responses to three or more questions (or a score of 3 or more) suggesting the presence of a probable opioid use disorder.
  units on a scale | 6.22 (1.36) | 6.04 (1.52) | 6.13 (1.44)
Severity of Opioid Use Disorder [Count of Participants; unit: Participants] — Measurement of the severity of opioid use disorder as indicated by the Structured Clinical Interview for DSM-5.
  Participants
    Mild | 8 | 13 | 21
    Moderate | 11 | 14 | 25
    Severe | 79 | 75 | 154

OUTCOME MEASURES:

1. Primary Outcome: Retention on Buprenorphine Treatment According to TimeLine Follow-Back - 3-months
Description: In this study, "retention on buprenorphine treatment" was defined as the time until a participant stopped taking their medication for 7 or more days in a row. This information was collected using a calendar recall method, the TimeLine Follow-Back (TLFB) measure at 3 months. The average number of days participants remained on buprenorphine before this happened was calculated, using the data collected at 3-month follow-up.
Time Frame: 3-months post enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 98 | 102
days | 81.1 (26.6) | 75.4 (32.3)

2. Secondary Outcome: Retention on Buprenorphine Treatment According to TimeLine Follow-Back - 12 Months
Description: In this study, "retention on buprenorphine treatment" was defined as the time until a participant stopped taking their medication for 7 or more days in a row. This information was collected using a calendar recall method, the TimeLine Follow-Back (TLFB) measure at 12 months. The average number of days participants remained on buprenorphine before this happened was calculated, using the data collected at 12-month follow-up.
Time Frame: 12-months post enrollment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 98 | 102
days | 252.1 (135.5) | 236.5 (148.9)

3. Secondary Outcome: Average Change in Self-reported Level of Pain Intensity on the Numerical Rating Scale for Pain Intensity (NRS-I) at 3-month Follow up (Compared to Baseline)
Description: Pain level will be measured using the Numerical Rating Scale for Pain Intensity (NRS-I), an 11-point numeric rating scale (0=no pain, 10= worst pain imaginable), which will be collected at the baseline enrollment assessment and 3-month follow-up. To calculate our measure, we subtracted each participant's score at 3-month assessment and subtracted it from their baseline score. We then averaged calculated average change in scores for each intervention group.
Time Frame: 3-months post enrollment
Population: Participants were not required to answer every survey question. Number of participants analyzed reflects number of participants who provided data for this survey question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 77 | 77
score on a scale | -0.7 (1.4) | -1.1 (2.2)

4. Secondary Outcome: Average Change in Self-Reported Level of Pain Related Functioning on the Brief Pain Inventory - Short Form (BPI) at 3-month Follow up (Compared to Baseline)
Description: Pain-related functioning will be measured using the pain interference subscale of the Brief Pain Inventory - Short Form (BPI), an 11-point numeric rating scale (0 = no pain/does not interfere, 10 = worst pain imaginable/completely interferes). For this study, an increase in pain-related functioning will be measured as a reduction in the pain interference scale scores over time. The BPI interference subscale measures how much pain has interfered with seven daily activities and will provide a current level of pain-related functioning (past 24-hours) at the 3-month follow-up. BPI pain interference will be calculated as the mean of the seven interference items. For each follow-up time point, the baseline value will be subtracted to obtain a change score.
Time Frame: 3-months post enrollment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 76
score on a scale | -0.3 (2.1) | -0.8 (2.2)

5. Secondary Outcome: Percent Days Abstinent From Substance Use on the TimeLine Follow-Back - 3-months
Description: Frequency of substance use will be measured using the TimeLine Follow-Back and will be collected at 3-month follow-up. During the administration, the participant will be asked to recall their alcohol and drug use utilizing a calendar-assisted structured interview that provides the participant with temporal cues to increase the accuracy of recall. At each follow-up, data will be collected for the entire period since the previous date of data collection. Percent days abstinent from substances (e.g. alcohol and drugs) will be used as the primary measure of substance use. Values shown are the treatment group average percent of days that participants were abstinent from substances after 3 months follow-up.
Time Frame: 3-months post enrollment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 85 | 86
percent of days | 76.7 (37.5) | 74.2 (37.8)

6. Secondary Outcome: Average Change in Self-reported Level of Pain Intensity on the Numerical Rating Scale for Pain Intensity (NRS-I) at 12-month Follow up (Compared to Baseline)
Description: Pain level will be measured using the Numerical Rating Scale for Pain Intensity (NRS-I), an 11-point numeric rating scale (0 = no pain, 10 = worst pain imaginable), which will be collected at the baseline enrollment assessment and the 12-month follow-up. For each follow-up time point, the baseline value will be subtracted to obtain a change score.
Time Frame: 12-months post enrollment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 66 | 68
score on a scale | -1.5 (2.2) | -1.9 (2.6)

7. Secondary Outcome: Average Change in Self-Reported Level of Pain Related Functioning on the Brief Pain Inventory - Short Form (BPI) at 12-month Follow up (Compared to Baseline)
Description: Pain-related functioning will be measured using the pain interference subscale of the Brief Pain Inventory - Short Form (BPI), an 11-point numeric rating scale (0 = no pain/does not interfere, 10 = worst pain imaginable/completely interferes). For this study, an increase in pain-related functioning will be measured as a reduction in the pain interference scale scores over time. The BPI interference subscale measures how much pain has interfered with seven daily activities and will provide a current level of pain-related functioning (past 24-hours) at the 12-month follow-up. BPI pain interference will be calculated as the mean of the seven interference items. For each follow-up time point, the baseline value will be subtracted to obtain a change score.
Time Frame: 12-months post enrollment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 62 | 67
score on a scale | -0.6 (2.9) | -0.9 (2.5)

8. Secondary Outcome: Percent Days Abstinent From Substance Use on the TimeLine Follow-Back - 12 Months
Description: Frequency of substance use will be measured using the TimeLine Follow-Back and will be collected at the 12-month follow-up. During the administration, the participant will be asked to recall their alcohol and drug use utilizing a calendar-assisted structured interview that provides the participant with temporal cues to increase the accuracy of recall. At each follow-up, data will be collected for the entire period since the previous date of data collection. Percent days abstinent from substances (e.g. alcohol and drugs) will be used as the primary measure of substance use. Values shown are the treatment group average percent of days that participants were abstinent from substances after 12 months follow-up.
Time Frame: 12-months post enrollment
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 68 | 73
percent of days | 74.7 (35.2) | 79.6 (32.0)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Psychosocial Pain Management (PPMI) | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 1/98 | 1/102
Serious Adverse Events (participants affected / at risk) | 20/98 | 16/102
Other Adverse Events (participants affected / at risk) | 10/98 | 7/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychosocial Pain Management (PPMI) (N=98) | Enhanced Usual Care (EUC) (N=102)
Hospitalization - psych (Psychiatric disorders) | 4 (5) | 4 (4) — Hospitalization due to psychiatric concerns
Hospitalization - general medical (General disorders) | 16 (28) | 13 (18) — General medical care for pain or injuries
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psychosocial Pain Management (PPMI) (N=98) | Enhanced Usual Care (EUC) (N=102)
Emergency Medical Visit (General disorders) | 3 (3) | 0 (0)
Car Accident (General disorders) | 1 (1) | 0 (0)
Detox (General disorders) | 1 (1) | 4 (4)
Residential Substance Use Treatment (General disorders) | 2 (2) | 5 (6)
Injury - Fall (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT04433975/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04433975/ICF_002.pdf